CLINICAL TRIAL: NCT02442128
Title: Using Fentanyl and Propofol for Tracheal Intubation During Sevoflurane Induction Without Muscle Relaxants in Children: a Randomized Prospective Study
Brief Title: Fentanyl and Propofol for Tracheal Intubation During Sevoflurane Induction Without Muscle Relaxants in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ashraf Arafat Abdelhalim, Assistant professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-14-1071
Record Dates: First submitted 2015-05-02; First posted 2015-05-13 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia Intubation Complication
Keywords: Fentany; intubation; sevoflurane; children; Propofol
MeSH Terms: interventions — Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group1 (Active Comparator): comparison of different dosages of drugs ( Fentanyl / Propofol), fentanyl 2 μg/kg and propofol 2 mg/kg Both test drugs will be made up to 10 ml with saline. fentanyl will be first administered intravenously over 30 s followed by propofol over 20 s.
  Interventions: Drug: propofol /Fentanyl; Drug: Fentanyl / propofol
- Group 2 (Active Comparator): comparison of different dosages of drug ( Fentanyl / Propofol) ,fentanyl 2 μg/kg and propofol 3 mg/kg. Both test drugs will be made up to 10 ml with saline. fentanyl will be first administered intravenously over 30 s followed by propofol over 20 s.
  Interventions: Drug: propofol /Fentanyl; Drug: Fentanyl / propofol

INTERVENTIONS:
Drug: propofol /Fentanyl — fentanyl 2 μg/kg and propofol 2 mg/kg Both test drugs will be made up to 10 ml with saline. fentanyl will be first administered intravenously over 30 s followed by propofol over 20 s.
  Other Names: Fentanyl; Diprivan
Drug: Fentanyl / propofol — fentanyl 2 μg/kg and propofol 3 mg/kg. Both test drugs will be made up to 10 ml with saline. fentanyl will be first administered intravenously over 30 s followed by propofol over 20 s.
  Other Names: Fentanyl; Diprivan

SUMMARY:
Several methods have been proposed to improve intubating conditions and minimize sevoflurane induction time during sevoflurane induction in children. These include clonidine premedication, [5] addition of nitrous oxide, [6] opioids, [7,8] or propofol [9].

Four Studies evaluated sevoflurane alone for intubation (9-12).Aim of this study: is to evaluate the effects of two different dose of propofol preceded by a fixed dose of fentanyl during sevoflurane induction on quality of tracheal intubation in children undergoing elective surgery.

DETAILED DESCRIPTION:
All patients fasted 6 h for solid food, but clear fluids will be given for up to 4 h pre- operatively. All patients will be pre-medicated with 0.3 mg/kg oral midazolam (maximum dose of 12 mg) 30 min before induction and EMLA cream will be applied to the dorsum of both hands 1 h prior to surgery. Children who refuse to take oral premedication will be excluded. One parent will be allowed to accompany the child into the pre-operative holding area. On arrival in the anesthetic room, baseline heart rate, pulse oximeter oxygen saturation and non-invasive blood pressure will be measured. A side-stream connector for the measurement of end-tidal sevoflurane concentration and end-tidal carbon dioxide will be introduced between the face mask and a Mapelson D breathing system.

* Anesthesia will be induced by a circle system using a vaporizer concentration of 6% sevoflurane in an oxygen flow of 6 L/min. After loss of consciousness and the eyelash reflex, sevoflurane concentration will be reduced to 3 % and intravenous access will be secured in all children using a 22-G cannula sited on the dorsum of a hand and the facemask ventilation will be then assisted using a 10 cm H2O inspiratory pressure at a ventilatory frequency of 16min. Once IV cannula is administered the inspired concentration of sevoflurane was decreased to 1% in oxygen.
* The investigating anesthetist will open a sealed envelope allocating the patient to one of two groups: Group 1 = fentanyl 2 μg/kg and propofol 2 mg/kg or Group 2 = fentanyl 2 μg/kg and propofol 3 mg/kg. Both test drugs will be made up to 10 ml with saline. In both groups, fentanyl will be first administered intravenously over 30 s followed by propofol over 20 s.
* Ninety seconds after administration of propofol, laryngoscopy and tracheal intubation with an appropriate sized non cuffed tube will be performed using a suitable sized Macintosh laryngoscope by a second an experienced unbiased anesthetist who enters the room and, unaware of the patient's randomization group. Intubating conditions will be evaluated as proposed by Viby-Mogensen and colleagues [9]. Five factors will be considered for assessment, jaw relaxation; ease of laryngoscopy; vocal cord position; coughing; and patient movement as excellent (1), good (2) or poor (3).
* Overall intubating conditions will be recorded as 'excellent' if all score 1, 'good' if any scored 2, and 'poor' if there will be any scores of 3. Intubation will not be attempted if the vocal cords is closed to avoid airway complications and any failure to intubate the trachea or prolonged coughing on intubation will be managed using suxamethonium or a non-depolarising muscle relaxant where clinically indicated.
* Following successful tracheal intubation, the study will be ended at this point, ventilation will be gently assisted and anesthesia will be maintained at the discretion of the anesthesiologist. In both groups HR, MAP and SPO2 will be measured immediately before the inhaled induction, after propofol administration, prior to intubation, immediately after intubation and at 2 and 5min min after intubation. Occurrence of bradycardia, hypotension or other significant complication will be recorded.
* The first investigating anesthetist is unblinded and responsible for preparing and administering all drugs. The second anesthetist will be blinded to drug allocation, intubate patients, record all parameters, and grade the airway conditions

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II patients, Undergoing elective ENT surgery

Exclusion Criteria:

* • History or examination suggested a potentially difficult intubation,

  * Significant respiratory disease or poorly controlled asthma,
  * gastrooesophageal reflux,
  * neurological or neuromuscular disease,
  * any condition that would preclude the use of this technique,
  * known sensitivity to the drugs used,
  * history or examination suggestive of cardiac illness,
  * history of respiratory tract infection in the previous 2 weeks,
  * history of malignant hyperthermia or other myopathy,
  * who refused to undergo an inhalational induction,
  * Children in whom i.v. access had already been established.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The incidence of excellent intubating conditions | during start of endotracheal intubation (10 seconds)
  Intubating conditions will be evaluated as proposed by Viby-Mogensen and colleagues . Five factors will be considered for assessment, jaw relaxation; ease of laryngoscopy; vocal cord position; coughing; and patient movement as excellent (1), good (2) or poor (3).
  Overall intubating conditions will be recorded as 'excellent' if all score 1, 'good' if any scored 2, and 'poor' if there will be any scores of 3. Intubation will not be attempted if the vocal cords is closed to avoid airway complications and any failure to intubate the trachea or prolonged coughing on intubation will be managed using suxamethonium or a non-depolarising muscle relaxant where clinically indicated.

SECONDARY OUTCOMES:
The hemodynamic response | 15 minutes
  . In both groups HR, MAP and SPO2 will be measured immediately before the inhaled induction, after propofol administration, prior to intubation, immediately after intubation and at 2 and 5min min after intubation. Occurrence of bradycardia, hypotension or other significant complication will be recorded.
The duration of intubation | during endotracheal intubation (30 seconds)
  time between the initial introduction of the laryngoscope and the final placement of the tracheal tube
number of intubation attempts | 5 minutes
  number of intubation attempts before successful intubation
occurrence of complication | 1 day
  bradycardia, hypotension , laryngeal spasm, desaturation, stridor or other significant complication will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf A Abdelhalim, MD, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided